CLINICAL TRIAL: NCT03402048
Title: Randomized Phase III Multicenter Trial of Customized Chemotherapy Versus Standard of Care for1st Line Treatment of Elderly Patients With Advanced Non-Small-Cell Lung Cancer
Brief Title: The EPIC Trial The Elderly Patient Individualized Chemotherapy Trial
Acronym: EPIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Prof. Silvia Novello, Principal Investigator, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-001194-81
Record Dates: First submitted 2014-11-17; First posted 2018-01-17 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Stage IV, NSCLC; Lung Neoplasms; Bronchial Neoplasms; Carcinoma, Bronchogenic; Lung Diseases; Neoplasms; Respiratory Tract Diseases; Respiratory Tract Neoplasms; Thoracic Neoplasms
Keywords: Lung Cancer; Elderly; First line; Customized chemotherapy; Pharmacogenomic-driven; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Bronchial Neoplasms; Carcinoma, Bronchogenic; Lung Diseases; Neoplasms; Respiratory Tract Diseases; Respiratory Tract Neoplasms; Thoracic Neoplasms | interventions — Carboplatin; Gemcitabine; Pemetrexed; Docetaxel; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control arm (Active Comparator): At discretion of the treating phisician. Common chemotherapic regimens include:
  Gemcitabine at 1000 or 1250 mg/m2 IV (in the vein) on day 1 and 8 of each 21 day cycle.
  Carboplatin at an AUC of 5 IV on day 1 of each 21 day cycle plus Gemcitabine at 1000 mg/m2 IV on Day 1 and 8 of each 21 day cycle.
  Carboplatin at an AUC of 5 IV on Day 1 of each 21 day cycle plus Pemetrexed 500mg/m2 on day 1 IV on Day 1 of each 21 day cycle.
  Vinorelbine 30 mg/m2 IV on day 1 and day 8 every 3 of each 21 day cycle.
  Number of Cycles: to a maximum of 6 cycles until progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Gemcitabine; Drug: Pemetrexed; Drug: Docetaxel; Drug: Vinorelbine
- experimental arm (Experimental): Treatment prescriptions will be based on gene analysis:
  * Carboplatin at an AUC of 6 IV (in the vein) on day 1 of each 21 day cycle.
  * Gemcitabine at 1000 mg/m2 IV on day 1 and 8 of each 21 day cycle.
  * Carboplatin at an AUC of 5 IV on day 1 of each 21 day cycle plus Gemcitabine at 1000 mg/m2 IV on Day 1 of each 21 day cycle.
  * Carboplatin at an AUC of 5 IV on Day 1 of each 21 day cycle plus Pemetrexed at 500 mg/m2 IV on Day 1 of each 21 day cycle.
  * Pemetrexed 500mg/m2 IV on Day 1 of each 21 day cycle.
  * Docetaxel 75 mg/m2 IV on Day 1 of each 21 day cycle. Or Vinorelbine 30 mg/m2 IV on day 1 and day 8 of each 21 day cycle.
  Number of Cycles: to a maximum of 6 cycles until progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Gemcitabine; Drug: Pemetrexed; Drug: Docetaxel; Drug: Vinorelbine

INTERVENTIONS:
Drug: Carboplatin
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Pemetrexed
  Other Names: Alimta
Drug: Docetaxel
  Other Names: Taxotere
Drug: Vinorelbine
  Other Names: Navelbine

SUMMARY:
This is a randomized phase III trial that will randomize elderly patients(70 years of age and older) who are not considered eligible for standard doublet or triplet regimens. In a 2:1 fashion, patients will be randomized to the customization arm or the standard arm, respectively. This trial will be offered to patients who are previously untreated for stage IV NSCLC.

The primary objective is to evaluate if chemotherapy selection based on histology and tumoral molecular determinants ERCC1, RRM1 and TS (arm A, the experimental arm) results in superior outcome in elderly patients with untreated, advanced NSCLC compared to standard of care treatments (arm B, the standard arm).

DETAILED DESCRIPTION:
The study population will consist of patients with histologically or cytologically proven stage IV NSCLC, who have not been previously treated with chemotherapy for stage IV and are either elderly (70 years of age and older). Patients must fulfill all the inclusion/exclusion criteria to be eligible.

Tissue will be obtained, and gene expression analysis will be performed at the University of Turin. The tissue sample used for this analysis will be obtained from the biopsy procedure performed as standard of care procedures during the patient's diagnosis and staging. Patients will be randomized to either Arm A: Experimental or Arm B: Standard of Care in a 2:1 fashion.

Tissue will be obtained for gene analysis for ALL patients. However, ONLY patients randomized to Arm A will receive the genetic analysis results. Genetic results will not be disclosed to the registering center for those patients randomized to Arm B: Standard of Care.

For patients randomized to Arm A: Experimental arm, the chemotherapy treatment prescription will be based on the gene analysis according to the protocol. For patients randomized to Arm B: Standard of Care arm, the chemotherapy treatment will be at the discretion of the care provider.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed NSCLC.

* Stage IV NSCLC by the AJCC Staging Manual 7th edition (2010).
* Measurable or evaluable disease by RECIST 1.1.
* Age equal or more than 70 years.
* Performance Status 0 or 1 (by ECOG criteria).
* Adequate bone marrow function.
* Signed informed consent document (ICD).
* Men with partners in the childbearing age group must use effective contraception.
* Previous surgery for NSCLC (more than 30 days before study registration) is allowed.
* Previous radiotherapy is allowed if: the time between completion of RT and initiation of study treatment is at least 7 days,the patient has fully recovered from all toxic effects, and at least one target lesion or evaluable disease is outside the radiation field.
* Previous chemotherapy is allowed if the last dose was administered equal to or greater than 12 months ago. This chemotherapy must have been given in an adjuvant or neoadjuvant mode prior to or after a curative intent surgical resection for a NSCLC. Patient should be previously untreated for metastatic disease.
* Patients with stable brain metastases will be allowed to enroll. Stable brain metastasis is defined as no progression of brain metastases 14 days after conclusion of definitive treatment as documented by a CT scan or MRI of the brain.

Exclusion Criteria:

* Prior systemic chemotherapy or immunotherapy for advanced NSCLC.
* Prior malignancies, except: cured non-melanoma skin cancer, curatively treated in situ carcinoma of the cervix, or any other curatively treated malignancy with no evidence of disease recurrence for at least 2 years.
* Presence of uncontrolled brain or leptomeningeal metastases.
* Peripheral neuropathy or hearing loss of neural origin equal to or greater than grade 2 by CTCAE v 4.0 except if due to trauma.
* Other serious illness or medical condition, including but not limited to: congestive heart failure;myocardial infarction within 6 months;significant neurologic or psychiatric disorders that would impact study participation as judged by the treating physician; infection requiring I.V. antibiotics; tuberculosis with ongoing therapy at study entry, superior vena cava syndrome, except if controlled with radiation, active peptic ulcer disease; unstable diabetes mellitus;any contraindication to high dose corticosteroid therapy such as herpes simplex, herpes zoster, hepatitis, or other disease.
* Hypercalcemia requiring therapeutic intervention.
* Clinically significant ascites and/or pericardial effusion.
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80.
* Concurrent treatment with other investigational drugs.
* Patients known to harbor sensitizing EGFR mutations in exons 18, 19 and 21. Patients with resistance mutation in exon 20 will be allowed to enroll i.e. T790M and D770. The rare patient who has both a resistance mutation and a sensitizing mutation at the diagnoses will be excluded in the protocol.
* Patients whose tissue submission is not of adequate size to perform molecular testing will be excluded.
* Patients known to have translocations of ALK will also be excluded; however, testing for ALK translocation prior to study entry is not mandated.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 567 (Estimated)
Dates: Start 2012-07; Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | from the date of randomization
  primary endpoint is OS (determined from the date of randomization).Assuming an exponential survival distribution for both treatment arms and a median survival time of 8 months in the control arm we anticipate to detect an improvement of three months in OS.

SECONDARY OUTCOMES:
Progression Free survival | at six months determined from the date of randomization
  PFS at 6 months (determined from the date of randomization). The anticipated 6-month PFS in arm B is approximately 25% and the goal in the experimental arm is to achieve a 32% improvement to 33%.

OTHER OUTCOMES:
AE and SAE (according to CTCAE version 4.0) | every week from the day 1 treatment until the end of treatment (up to 18 weeks)
  adverse events and serious adverse events as a measure of safety and tolerability
Rate of successfully conducted gene expression analysis in patients that have signed the informed consent document | up to10 business days of submission of the tumor specimen
  Rate of successfully conducted gene expression analysis in patients that have signed the informed consent document

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Novello, MD, PhD, Principal Investigator — University of Turin, Italy; Giorgio Vittorio Scagliotti, MD, PhD, Principal Investigator — Univerisity of Turin; Tiziana Vavalà, MD, Principal Investigator — University of Turin, Italy
Locations (28):
- Italy (28):
  - IRCSSIstituto Scientifico Romagnolo per lo studio e la cura dei tumori IRST, Meldola, Forlì
  - Istituto Nazionale Tumori, Aviano, Pordenone
  - Ospedale di Faenza, Faenza, Ravenna
  - Ospedale di Lugo, Lugo, Ravenna
  - AUSL Rimini-Oncologia Medica Cattolica, Cattolica, Rimini
  - AOU San Luigi Gonzaga, Department of Oncology, University of Turin, Orbassano, Turin
  - Ospedale Giovanni Paolo II, Bari
  - AO Cannizzaro, Catania
  - AOU Santa Croce e Carle, Cuneo
  - Azienda Ospedaliera Careggi, Florence
  - Istituto Nazionale per la Ricerca sul Cancro, Genova
  - Ospedale Galliera, Genova
  - Azienda Ospedaliera Fatebenefratelli, Milan
  - Ospedale S. Raffaele, Milan
  - AO San Gerardo, Monza
  - Istituto Oncologico Veneto, Padua
  - Ospedale Santa MAria della Misericordia, Perugia
  - Ospedale S MAria delle Croci, Ravenna
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - AUSL Rimini-Oncologia medica, Rimini
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Ospedale S. Giovanni Addolorata, Roma
  - Policlinico Umberto I- Università la Sapienza, Roma
  - AOU Sassari, Sassari
  - Azienda Ospedaliera Sondalo, Sondalo
  - Ospedale Santa Chiara, Trento
  - AOU S.M. Misericordia, Udine
  - AOU Verona, Verona